CLINICAL TRIAL: NCT02517242
Title: Syringes Replacement for Insulin Application for Pens Device in a Population of Elderly Patients With Type 2 Diabetes: Multifactorial Intervention to Improve Glycemic controlCONTROL
Brief Title: Syringes Replacement for Insulin Application for Pens Device in a Population of Elderly Patients With Type 2 Diabetes: Multifactorial Intervention to Improve Glycemic Control
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Principal Investigator, Ticiana da Costa Rodrigues, Professor of Medicine, Hospital de Clinicas de Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13-0485
Record Dates: First submitted 2015-08-03; First posted 2015-08-06 (Estimated); Last update posted 2015-08-06 (Estimated); Status verified 2015-08

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus | interventions — Syringes; Blood Glucose

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pens Device (Experimental): All patients will receive pens device, insulin, blood glucose monitor, lancet tapes, capillary blood glucose tests (3 tests/day). All will be evaluated monthly for six months
  Interventions: Device: Pens Device; Other: Monitoring capillary blood glucose with blood glucose monitor, lancet tapes and capillary blood glucose tests (3 tests/day)
- Syringe (Active Comparator): All patients will receive syringe to insulin, insulin, blood glucose monitor, lancet tapes, capillary blood glucose tests (3 tests/day). All will be evaluated monthly for six months
  Interventions: Device: Syringe; Other: Monitoring capillary blood glucose with blood glucose monitor, lancet tapes and capillary blood glucose tests (3 tests/day)

INTERVENTIONS:
Device: Pens Device
  Arms: Pens Device
Device: Syringe
  Arms: Syringe
Other: Monitoring capillary blood glucose with blood glucose monitor, lancet tapes and capillary blood glucose tests (3 tests/day)

SUMMARY:
This is a prospective, intervention, randomized, phase IV study. Patients will be included with 60 years or older, both sexes, with HbA1c >8.5% using oral antidiabetics agents and insulin and then we will be randomized by use syringe or pens device to use insulin NPH and regular. All patients will receive a blood glucose monitor, lancet tapes, capillary blood glucose tests (3 tests/day). HbA1c will be measured at baseline, 3 and 6 months. Patients will see monthly.

ELIGIBILITY:
Inclusion Criteria:

* Sixty years or older
* Diabetes type 2 with Glycated Hemoglobin higher than 8.5%
* Using or necessity to use insulin
* Using syringe to insulin
* Using at least one oral antidiabetic
* Accept to participate

Exclusion Criteria:

* Glomerular Filtration Rate lower than 30
* Considering unfit for self administration of insulin

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2015-05; Primary Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Glycated Hemoglobin | reduction compared to baseline values at six months
  reduction compared to baseline values

SECONDARY OUTCOMES:
Blood Pressure | reduction compared to baseline values at six months
  Monthly measurements are made
adherence | reduction compared to baseline values at six months
  Monthly measurements are made
Number of pills, antidiabetics drugs and antihypertensives drugs | reduction compared to baseline values at six months
  Monthly measurements are made
Number of hypoglycemias | reduction compared to baseline values at six months
  Monthly measurements are made
Presence of severe hypoglycemias | reduction of the number of patients with this outcome compared to baseline values at six months
  Monthly measurements are made
Presence of nocturnal hypoglycemias | reduction of the number of patients with this outcome compared to baseline values at six months
  Monthly measurements are made
Presence of asyntomatic hypoglycemias | reduction of the number of patients with this outcome compared to baseline values at six months
  Monthly measurements are made

CONTACTS AND LOCATIONS:
Overall Officials: Ticiana da Costa Rodrigues, Principal Investigator — Hospital de Clínicas de Porto Alegre
Locations (1):
- Rafael Vaz Machry, Porto Alegre, Rio Grande do Sul, Brazil

REFERENCES:
- [Derived] Machry RV, Cipriani GF, Pedroso HU, Nunes RR, Pires TLS, Ferreira R, Vescovi B, de Moura GP, Rodrigues TC. Pens versus syringes to deliver insulin among elderly patients with type 2 diabetes: a randomized controlled clinical trial. Diabetol Metab Syndr. 2021 Jun 12;13(1):64. doi: 10.1186/s13098-021-00675-y. PMID 34118981